CLINICAL TRIAL: NCT04516681
Title: Vitamin C Intravenously With Chemotherapy and Adebrelimab in Metastatic Colorectal Cancer With High Expresison Level of GLUT3
Brief Title: Combination of IV Ascorbic Acid and Adebrelimab in Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, Dr., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin C-GLUT3-2020
Record Dates: First submitted 2020-08-12; First posted 2020-08-18 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Vitamin C; GLUT3
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ascorbic Acid; Folfox protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Ascorbic Acid with Adebrelimab and chemotherapy group (Experimental): Ascorbic Acid with Adebrelimab and FOLFOX ± bevacizumab. Ascorbic Acid (1.5g/kg/day, D1-3) every 2 weeks
  Interventions: Drug: Ascorbic acid; Drug: FOLFOX Protocol; Drug: Adebrelimab
- Chemotherapy alone group (Active Comparator): standard FOLFOX treatment
  Interventions: Drug: FOLFOX Protocol

INTERVENTIONS:
Drug: Ascorbic acid — 1.5g/kg/day, D1-3, every 2 weeks
  Other Names: Vitamin C
  Arms: Combined Ascorbic Acid with Adebrelimab and chemotherapy group
Drug: FOLFOX Protocol — Oxaliplatin 130 mg/m² d1 concurrent with Leucovorin 400 mg/m², followed by Oxaliplatin 85 mg/m² d1 followed by Bolus 5FU 400 mg/m² , followed by Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks with or without bevacizumab 5mg/kg, every 2 weeks
  Other Names: FOLFOX+/- bevacizumab
Drug: Adebrelimab — 20mg/Kg intravenously every 3 weeks
  Arms: Combined Ascorbic Acid with Adebrelimab and chemotherapy group

SUMMARY:
Previous preclinical study has shown that high levels of ascorbic acid (AA) possesses the ability to kill human colorectal cancer cells and high expression of GLUT3 will augment the efficacy of AA. To date, no previous studies have investigated the combination of therapeutic role of AA and PD-L1 antibody in metastatic colorectal cancer with high expression of GLUT3. This protocol is a randomized controlled study of AA infusions combined with Adebrelimab and FOLFOX +/- bevacizumab versus treatment with FOLFOX +/- bevacizumab alone in metastatic colorectal cancer patients with high expression of GLUT3.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years, ≤75 years; Histologically proven peritoneal metastatic adenocarcinoma of colorectal cancer, unresectable metastatic disease; IHC confirmed strong positive GLUT3; measurable disease; Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1; Life expectancy of at least 12 weeks; ANC ≥1,500/mm3; Hemoglobin > 8g/dL; platelet ≥ 100,000/mm3; Laboratory at baseline evaluation for inclusion in the study: creatinine ≤1.5X upper limit [if the creatinine is elevated, but ≤1.5X the ULN, a 24 hour creatinine clearance will be obtained, Creatinine clearance > 50 mL/min (calculated according to Cockroft and Gault)]; Transaminase (AST/ALT) ≤2.5X upper limit of normal and bilirubin levels ≤1.5X upper limit of normal without liver metastasis; Transaminase (AST/ALT) ≤5X upper limit of normal and bilirubin levels ≤1.5X upper limit of normal with liver metastasis; Written informed consent

Exclusion Criteria:

* Prior treatment for metastatic disease (adjuvant therapy with fluoropyrimidines +/-oxaliplatin based regimens allowed if stopped 12 months prior to registration on study); Surgery (excluding diagnostic biopsy) or irradiation within 3 weeks prior to study entry; Administration of any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment; Concurrent chronic systemic immune therapy, chemotherapy, radiation therapy (palliative radiation therapy allowed) or hormone therapy not indicated in the study protocol; Brain metastasis (known or suspected); Pregnant or lactating women; Other uncontrolled concomitant illness, including serious uncontrolled intercurrent infection; Known allergy or any other adverse reaction to any of the drugs or to any related compound; Previous (within 5 years) or concurrent malignancies at other sites with the exception of surgically cured or adequately treated carcinoma in-situ of the cervix and basal cell carcinoma of the skin; Patients with low or moderate expression of GLUT3.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 5 years
  To utilize CT or MRI scans to assess overall tumor response rate (complete and partial response) in subjects with peritoneal metastatic colorectal cancer treated with the combination of ascorbic acid and FOLFOXIRI +/- bevacizumab versus treatment with FOLFOXIRI +/- bevacizumab alone

SECONDARY OUTCOMES:
Progression Free Survival | up to 5 years
  Time-to-event outcome measure (initial disease progression) measured in days from cycle 1 day 1 to day of first progression as defined by RECIST1.1 criteria from NCI
Overall Survival | up to 5 years
  Time to event outcome measure (death), measured in days from cycle 1 day 1

CONTACTS AND LOCATIONS:
Overall Officials: Guoxiang Cai, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan university shanghai cancer center, Shanhai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No